CLINICAL TRIAL: NCT01256970
Title: The Study of Polycystic Ovary Syndrome (PCOS) and Questionnaire
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Ming-I Hsu, Attending Doctor, Taipei Medical University WanFang Hospital
Other Study IDs: WFH-PCOS-99075
Record Dates: First submitted 2010-12-07; First posted 2010-12-09 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Polycystic Ovary Syndrome.: Polycystic ovary syndrome was diagnosed according to the 2003 Rotterdam criteria, which require a minimum of two of the following three criteria: PCOM, chronic anovulation and hyperandrogenism.
- Normal Control: Normal control women were women who did not present with any of three PCOS criteria.

SUMMARY:
Polycystic ovary syndrome (PCOS) is an extremely common disorder in women of reproductive age. Diagnosis of PCOS is principally based on clinical and physical findings. Diagnostic criteria and PCOS definitions used by clinicians and researchers are almost as heterogeneous as the syndrome. This first part of study is determine whether genetic polymorphisms influence hormonal and metabolic characteristics in Taiwanese patients with PCOS and controls. Furthermore, women with PCOS were reported with high risk of cardiovascular disease, the investigators planned to calculate the difference of carotid intima-media thickness (IMT) and B-type natriuretic peptide (BNP) between women with PCOS and normal control to determine the premature atherosclerosis of women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* women at reproductive age
* women with PCOS and women without PCOS

Exclusion Criteria:

* young women who had their menarche less than 3 years
* women older than 45 years old, Amenorrhea of menopause, hyperglycemia, hyperthyroidism, hypothyroidism, heart failure, lung failure, renal failure, anemia, dystrophy, gonitis

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Polycystic Ovary Syndrome(PCOS)
Sampling Method: Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2010-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Obesity is the predominant predictor of impaired glucose tolerance and metabolic disturbance in polycystic ovary syndrome. | Prospectively study in University teaching hospital from 31 August 2010 to 31 August 2011.
  To evaluate the contribution to glucose intolerance and metabolic syndrome of obesity combined with the diagnostic criteria of polycystic ovary syndrome (PCOS).

CONTACTS AND LOCATIONS:
Overall Officials: Ming-I Hsu, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University-WanFang Hospital, Taipei, Taiwan